CLINICAL TRIAL: NCT00784940
Title: A Randomised, Double-Blind Trial to Assess the Effects on Bone Mineral Density and Metabolism of Arimidex Alone, Nolvadex Alone, or Arimidex and Nolvadex in Combination, (in Comparison to a Control Group) When Used as Adjuvant Treatment for Breast Cancer in Postmenopausal Women
Brief Title: ATAC - Bone Density Sub-Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar, Medical Science Director, Arimidex and Faslodex, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1033ID/0029; D5392C01985
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Bone Density
MeSH Terms: interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Arimidex 1mg + Nolvadex placebo
  Interventions: Drug: Anastrozole
- 2 (Active Comparator): Arimidex placebo + Nolvadex 20mg
  Interventions: Drug: Anastrozole; Drug: Tamoxifen
- 3 (Active Comparator): Arimidex 1mg + Nolvadex 20mg
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — 1mg, orally, once daily
  Other Names: Arimidex
  Arms: 1; 2
Drug: Tamoxifen — 20mg, orally, once daily
  Other Names: Nolvadex
  Arms: 2; 3

SUMMARY:
To assess and quantify the changes in bone mineral density between the ARIMIDEX and ARIMIDEX plus NOLVADEX groups when compared to the NOLVADEX alone treatment group whilst receiving trial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for entry into the main ATAC trial 1033IL/0029
* Women defined as post-menopausal
* Patients with histologically proven operable invasive breast cancer
* Who following primary surgery have a good prognosis and would be ethically suitable to remain untreated

Exclusion Criteria:

* Excluded from entry into the main ATAC trial (1033IL/0029)
* Patients who have received hormone replacement therapy within the previous 12 months prior to randomisation
* Patients who have received bisphosphonate therapy within the previous 12 months prior to randomisation
* Patients who have had a bone fracture within the previous 6 months prior to randomisation

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 1998-06; Primary Completion 2005-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time to withdrawal
Time to recurrence